CLINICAL TRIAL: NCT06892418
Title: A Clinical Study on the Effects of Ketoflex 12/3 Diet on Motor and Non-Motor Symptoms in Patients With Parkinson's Disease
Brief Title: Impact of Ketoflex 12/3 Diet on Parkinson's Disease Symptoms: A Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Prof. Lutfu Hanoglu, MD, Professor.MD.PhD, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PD23992
Record Dates: First submitted 2025-03-21; First posted 2025-03-24 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Parkinson's Disease; Parkinson
Keywords: Parkinson's Disease; Ketogenic Diet; Intermittent Fasting; Ketoflex 12/3; Neurodegenerative Disorders
MeSH Terms: conditions — Parkinson Disease; Intermittent Fasting; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketoflex 12/3 Diet Group (Experimental): A plant-based ketogenic diet combined with intermittent fasting (12/3)
  Interventions: Behavioral: Ketoflex 12/3 Diet
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Ketoflex 12/3 Diet — A plant-based ketogenic diet combined with intermittent fasting (12/3)
  Arms: Ketoflex 12/3 Diet Group

SUMMARY:
This study aims to investigate the effects of the Ketoflex 12/3 diet on motor and non-motor symptoms in patients with Parkinson's disease. Participants will follow the Ketoflex 12/3 dietary regimen, and their cognitive function, motor symptoms, sleep patterns, gastrointestinal health, and overall well-being will be assessed through standardized clinical scales. The study will help determine whether a plant-based ketogenic diet combined with intermittent fasting can have a beneficial impact on Parkinson's disease progression.

DETAILED DESCRIPTION:
Parkinson's disease is a progressive neurodegenerative disorder characterized by motor and non-motor symptoms. Emerging evidence suggests that dietary interventions, particularly ketogenic diets and intermittent fasting, may play a role in neuroprotection and symptom management. This study investigates the effects of the Ketoflex 12/3 diet, a plant-based ketogenic dietary approach combined with intermittent fasting, on Parkinson's disease progression. Clinical assessments will include Unified Parkinson's Disease Rating Scale (UPDRS), Mini-Mental State Examination (MMSE), depression and anxiety scales, sleep quality assessments, and gastrointestinal health evaluations. The study aims to provide new insights into the potential benefits of metabolic-based nutritional interventions in Parkinson's disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's disease
* Age between 40-85 years
* Native Turkish speakers
* Able to comply with the study protocol

Exclusion Criteria:

* History of alcohol or substance dependence
* Diagnosis of chronic renal failure
* Presence of neuromuscular disorders
* Having amalgam dental fillings and/or failure to remove them according to the SMART protocol
* Severe vitamin deficiencies that have not been corrected prior to the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Motor Symptoms as Measured by the Unified Parkinson's Disease Rating Scale (UPDRS) | Baseline and 6 months
  The Unified Parkinson's Disease Rating Scale (UPDRS) is used to evaluate the severity of motor symptoms in Parkinson's disease. Scores range from 0 to 108 for the motor section, with higher scores indicating worse motor impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medipol Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
At this time, no final decision has been made regarding individual participant data (IPD) sharing. Future data-sharing plans will be considered in accordance with institutional policies, ethical guidelines, and publication requirements